CLINICAL TRIAL: NCT00701363
Title: A Prospective, International, Multi-centric, Open-label Study to Assess the Efficacy of an Extended Injection Interval Schedule of Lanreotide Autogel 120 mg in Acromegalic Subjects Who Are Biochemically Controlled on the Long Term Treatment With Octreotide LAR 10 or 20 mg
Brief Title: Study to Assess the Efficacy of an Extended Injection Interval Schedule of Lanreotide Autogel in Acromegalic Subjects
Acronym: LEAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-38-52030-214; 2007-005838-37 (EudraCT Number)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

ARMS (1):
- Lanreotide Autogel 120 mg (Experimental)
  Interventions: Drug: Lanreotide Autogel 120 mg

INTERVENTIONS:
Drug: Lanreotide Autogel 120 mg — 120mg, injections every 6 weeks, then depending on IGF-1 results at Week 24

SUMMARY:
The purpose of the study is to assess the efficacy of an extended injection interval schedule of lanreotide Autogel 120 mg in acromegalic subjects who are biochemically controlled on long term treatment with octreotide LAR 10 or 20 mg

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written informed consent prior to any study-related procedures
* The subject is male or female and is over 18 years of age
* The subject must have had documentation supporting the diagnosis of acromegaly, based on elevated IGF-1 and/or GH levels
* The subject has been receiving octreotide LAR (10 or 20 mg) treatment for at least six months and is biochemically controlled. Control is defined as normal (age and sex adjusted) IGF 1 levels for two consecutive measurements (at least two months apart) preceding study entry
* If the subject is receiving dopamine agonist therapy, treatment should be stable for at least four months, and no change in their dopamine-agonist medication is expected during the entire study period

Exclusion Criteria:

* The subject has received radiation therapy to the pituitary gland before study entry
* The subject has a history of hypersensitivity to lanreotide or drugs with a similar chemical structure
* The subject has received a growth hormone receptor antagonist (pegvisomant) therapy within three months before study entry
* The subject has undergone treatment with any other investigational drug in the 30 days before study entry or is scheduled to receive an investigational drug, other than lanreotide 120 mg, during the course of the study
* The subject has received any unlicensed drug within the 30 days prior to the baseline visit or is scheduled to receive an unlicensed drug during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (44):
- Brazil (2):
  - Universidade Federal do Rio de Janeiro - Department of Internal Medicine - Section of Endocrinology - Neuroendocrine Research Center, Rio de Janeiro
  - Hospital das Clínicas de São Paulo - Internal Medicine - Neuroendocrine Unit - Division of Endocrinology and Metabolism, São Paulo
- Denmark (3):
  - Arhus University Hospital - Department of Medicinsk AVd M, Arhus C
  - Righospitalet - University Department of Endocrinology & Internal Medicine P, Copenhagen
  - Odense University Hospital - Department of Endocrinology, Odense C
- Finland (2):
  - Helsinki University Central Hospital - (HUCH) Division of Endocrinology - Department of Medicine, Helsinki
  - Kuopio University Hospital - Department of Medicine, Internal Medicine/Endocrinology and Diabetology Division, Kuopio
- France (15):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Hôpital Avicenne - Bâtiment Madeleine Breis, Bobigny
  - Hôpital Neurologique - Pierre Wertheimer, Bron
  - Hôpital du Bocage Sud - Service d'Endocrinologie, Dijon
  - CH La Rochelle - Hopital Saint Louis - Service de Médecine interne - Endocrinologie - Maladies Métaboliques- Nutrition, La Rochelle
  - Hôpital Du Cluzeau - Service de Médecine B, Limoges
  - Hôpital Archet 1 - Service d'Endocrinologie, Nice
  - CHU de Nîmes - Hôpital Caremeau, Nîmes
  - Hôpital Lariboisière - Service Médecine Interne - Endocrinologie - Nutrition, Paris
  - Hopital Pitié-Salpêtrière - Service d'Endocrinologie, Paris
  - Hôpital Cochin - Saint-Vincent-de-Paul - La-Roche-Guyon, Paris
  - Hôpital Haut Lévêque - Unité de soins normalisés, Pessac
  - Hôpital Robert Debré, Reims
  - Hôpital de Hautepierre, Service de Médecine Interne et Nutrition, Strasbourg
  - CHU de Tours - Hopital Bretonneau - Service Endocrinologie-Diabétologie Medecine B, Tours
- Greece (4):
  - Evangelismos Hospital - Department of Endocrinology, Athens
  - Polykliniki Hospital - Department of Endocrinology, Athens
  - Metaxa Hospital - Department of Endocrinology, Piraeus
  - B IKA Panagia Hospital - Department of Endocrinology, Thessaloniki
- P. Stradins Clinical University Hospital - Department of Endocrinology, Riga, Latvia
- Netherlands (2):
  - Erasmus Medical Centre - Department of Endocrinology, Rotterdam
  - UMC Utrecht - Department of Endocrinology, Heidelberglaan 100, Utrecht
- Department of Medicine, Haukeland Hospital Jonas Lies, Bergen, Norway
- Poland (3):
  - Swietorkryskie Centrum Onkologii, UL. Artwinskiego 3 - Department of endocrinology and Nuclear Medecine, Kielce
  - University Hospital in Krakow, Dept. of Endocrinology, Kopernika Str. 17, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Ul. Pasteura 4, Wroclaw
- University of Medicine and Pharmacy Iuliu Hatieganu, Cluj-Napoca, Romania
- Russia (2):
  - Federal State Institution "Endocrinology Research Centre - Federal agency of high-tech medical care" - Neuroendocrinology & Osteopathy Department, Moscow
  - I.M. Sechenov Moscow Medical Academy - Endocrinology Department, Moscow
- Serbia (2):
  - Clinical Centre of Serbia - Institute for Endocrinology, Diabetes and Metabolic Diseases, - Dr Subotica Street n°13, Belgrade
  - Clinic for Endocrinology, Diabetes and Metabolic Disorders, Clinical Center of Vojvodina, Hajduk Veljkova 3-9, Novi Sad
- South Korea (3):
  - Seoul National University hospital, 28 Yongon-dong Chongno-gu, Seoul
  - Yonsei University Severance Hospital - Department of Endocrinology and Metabolism, Seoul
  - Sungkyunkwan University Samsung Medical Center, Seoul
- Sweden (3):
  - EM-Kliniken, Universitetssjukhuset, Linköping
  - Skane University Hospital, Department of Endocrinology, Lund
  - Karolinska University Hospital, Dpt of Endocrinology, Metabolism & Diabetology, Solna, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiation date: 06-Oct-2008. Study completion date: 20-May-2013. Screened subjects were 128 and screen failure subjects were 4. Subjects treated were 124 and subjects withdrawn early were 17. Subjects completed the study were 107.
Groups:
- Phase 1: Lanreotide Autogel 120 mg: Subjects in phase 1 received 5 injections of Lanreotide Autogel 120 mg subcutaneously (SC) at baseline and weeks 6, 12, 18 and 24. Baseline and week 24 injections were administered in the investigational centre, whereas the patient could receive weeks 6, 12 and 18 injections at home as part of the subject's normal medical care, completing details of the injection in the diary cards provided.
- Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks: Subjects with IGF-1 levels >100% to ≤130% of ULN at week 24 were assigned to group A. These subjects received 5 injections of Lanreotide Autogel 120 mg at 4-week intervals from week 24 up to week 48.
- Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks: Subjects with IGF-1 levels >50% to ≤100% of ULN at week 24 were assigned to group B. These subjects received 3 injections of Lanreotide Autogel 120 mg at 6-week intervals from week 24 up to week 48.
- Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks: Subjects with IGF-1 levels ≤50% of ULN at week 24 were assigned to group C. These subjects received 2 injections of Lanreotide Autogel 120 mg at 8-week intervals from week 24 up to week 48.
Period: Screening (Pre-assignment) Phase
Arm/Group | Phase 1: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Started | 128 | 0 | 0 | 0
Completed | 124 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Does not meet entry Criteria | 4 | 0 | 0 | 0
Period: Treatment Phase 1
Arm/Group | Phase 1: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Started | 124 | 0 | 0 | 0
Completed | 109 | 0 | 0 | 0
Not Completed | 15 | 0 | 0 | 0
Not completed — Does not meet entry Criteria | 1 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Period: Treatment Phase 2
Arm/Group | Phase 1: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Started | 0 | 13 | 70 | 26
Completed | 0 | 13 | 68 | 26
Not Completed | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1: 15 subjects participated only in phase 1 and did not enter in phase 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks | Total
Number analyzed (Participants) | 15 | 13 | 70 | 26 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (15.3) | 55.0 (10.1) | 53.2 (10.4) | 57.0 (9.8) | 55.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 41 | 20 | 78
  Male | 6 | 5 | 29 | 6 | 46
Region of Enrollment [Number; unit: participants]
  Russian Federation | 1 | 3 | 12 | 4 | 20
  Korea, Republic of | 2 | 4 | 7 | 4 | 17
  Brazil | 2 | 0 | 12 | 1 | 15
  Serbia | 2 | 3 | 8 | 2 | 15
  France | 1 | 0 | 9 | 4 | 14
  Poland | 1 | 1 | 8 | 2 | 12
  Latvia | 1 | 0 | 7 | 2 | 10
  Greece | 2 | 0 | 3 | 4 | 9
  Sweden | 1 | 0 | 3 | 0 | 4
  Finland | 1 | 1 | 0 | 1 | 3
  Denmark | 0 | 0 | 0 | 2 | 2
  Norway | 1 | 0 | 0 | 0 | 1
  Romania | 0 | 0 | 1 | 0 | 1
  Netherlands | 0 | 1 | 0 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (2.9) | 29.2 (4.1) | 29.5 (6.5) | 27.0 (4.3) | 28.8 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Having Maintained Their Injection Interval Schedule of Six Weeks or Increased Their Injection Interval to Eight Weeks Whilst Keeping Their Normalised Insulin Growth Factor (IGF-1) Levels (Age and Sex Adjusted)
Description: A subject was responder if he maintained his injection interval schedule of 6 weeks or increased his injection interval to eight weeks whilst keeping his normalised IGF-1 level (age and sex adjusted) at the end of the study (Week 48)
Time Frame: At week 48 (End of Study)
Population: Intention to Treat (ITT) population: All patients having received ≥1 study drug dose. Modified ITT (MITT) population: All subjects in the ITT population for whom group allocation was performed (included in Phase 2).
  n = Number of subjects at the visit
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 124
Percentage of subjects
  Intention-to-Treat (n=124) | 75.8 [68.3 to 83.3]
  Modified Intention-to-Treat (n=109) | 86.2 [79.8 to 92.7]

2. Secondary Outcome: Percentage of Subjects With Normalised IGF-1 Levels (Age and Sex Adjusted)
Description: The criterion for a subject is satisfied if he has a normalised IGF-1 level (age and sex adjusted) at week 24.
Time Frame: At week 24
Population: ITT population. n = Number of subjects at the visit.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 124
Percentage of subjects
  Intention-to-Treat (n=124) | 88.7 [83.1 to 94.3]
  Modified Intention-to-Treat (n=109) | 100 [100 to 100]

3. Secondary Outcome: Percentage of Subjects Having Maintained an Injection Interval of Six Weeks or Increasing Their Injection Interval to Eight Weeks
Description: The criterion for a subject is satisfied if he maintained an injection interval of six weeks or increasing his injection interval to eight weeks during Phase 2 of the study.
Time Frame: During phase 2 of the study (up to week 48)
Population: ITT population. n = Number of subjects at the visit.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 124
Percentage of subjects
  Intention-to-Treat (n=124) | 78.2 [71.0 to 85.5]
  Modified Intention-to-Treat (n=109) | 88.1 [82.0 to 94.2]

4. Secondary Outcome: Percentage of Subjects Who Extend Their Injection Interval to Eight Weeks During Phase 2 of the Study, Whilst Maintaining Normalised IGF-1 Levels
Description: The criterion for a subject is satisfied if he extended his injection interval to eight weeks during Phase 2 of the study, whilst maintaining normalised IGF-1 levels at Week 48.
Time Frame: At week 48
Population: ITT population. n = Number of subjects at the visit.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 124
Percentage of subjects
  Intention-to-Treat (n=124) | 20.2 [13.1 to 27.2]
  Modified Intention-to-Treat (n=109) | 22.9 [15.0 to 30.8]

5. Secondary Outcome: Mean Change From Baseline in IGF-1 Values [Expressed as % of Upper Limit of Normal (ULN)], Overall and by Injection Interval
Description: IGF-1 change from Baseline to Week 48 = Mean IGF-1 level at Week 48 - Mean IGF-1 level at Baseline
Time Frame: Baseline (visit 1) and week 48
Population: MITT population. One subject (Group B) had missing IGF-1 value at Week 48. One subject (Group A) had missing IGF-1 value at Baseline.
Measure: Mean (Standard Deviation); unit: Percentage of ULN
Arm/Group | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Number analyzed (Participants) | 12 | 67 | 25
Percentage of ULN | -1.70 (18.55) | 5.74 (30.48) | -4.33 (28.14)
Statistical Analysis 1: Comparison: Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks vs Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks; One subject (Group B) had missing IGF-1 value at Week 48. One subject (Group A) had missing IGF-1 value at Baseline; Test type: Superiority or Other; p = 0.0013, ANCOVA
Statistical Analysis 2: Comparison: Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks vs Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks vs Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks; Test type: Superiority or Other; p < 0.0001, ANCOVA

6. Secondary Outcome: Treatment Group (A, B or C) Mean Baseline IGF-1 Levels (Expressed as % of ULN) in Subjects Who Maintained Normalised IGF-1 Values at Week 48. Comparisons Will be Made as Follows: A Versus B, A Versus C, A Versus (B+C) and B Versus C
Time Frame: Baseline (visit 1)
Population: MITT population.
  One subject in Group A had missing IGF-1 value at baseline. One subject in Group B had missing IGF-1 value at week 48 and two subjects did not attend week 48 (early withdrawal). One subject in Group C had missing IGF-1 value at week 48.
Measure: Mean (95% Confidence Interval); unit: Percentage of ULN
Arm/Group | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Number analyzed (Participants) | 12 | 67 | 25
Percentage of ULN | 98.69 [89.4 to 108.0] | 67.75 [60.4 to 75.1] | 51.30 [41.1 to 61.5]
Statistical Analysis 1: Comparison: Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks vs Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks; Test type: Superiority or Other; p = 0.0009, t-test, 2 sided
Statistical Analysis 2: Comparison: Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks vs Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks vs Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks vs Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks vs Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.0170, t-test, 2 sided

7. Secondary Outcome: Mean Baseline IGF-1 Levels (Expressed as % of ULN) in All Groups (A, B and C) Versus Mean Baseline IGF-1 Levels (Expressed as % of ULN) in Subjects With Uncontrolled IGF-1 Levels at Week 24
Time Frame: Baseline (visit 1)
Population: ITT population. n = Number of subjects at the visit.
  These subjects entered in phase 2
  One subject was not included in this analysis because IGF-1 was lower than 130% at week 24 but not in the second phase and one subject in group A had missing IGF-1 value at baseline.
Measure: Mean (95% Confidence Interval); unit: Percentage of ULN
Arm/Group | Overall Study
Number analyzed (Participants) | 122
Percentage of ULN
  Uncontrolled IGF-1 levels at Week 24 (n=14) | 95.92 [50.3 to 141.5]
  Normalized IGF-1 levels at Week 24 (A+B+C) (n=108) | 67.49 [61.8 to 73.2]
  Difference in Mean Baseline | 28.43 [6.83 to 50.03]
Statistical Analysis 1: Comparison: Overall Study; Difference in baseline IGF-1 levels between 108 subjects with normalized IGF-1 levels at week 24 (A+B+C) and 14 subjects with uncontrolled IGF-1 levels at week 24; Test type: Superiority or Other; p = 0.0103, t-test, 2 sided

8. Secondary Outcome: Symptoms of Acromegaly (Headache, Excessive Perspiration, Fatigue, Soft Tissue Swelling and Arthralgia)
Description: Acromegaly symptoms were assessed by the patients using the Patient Assessed Acromegaly Symptom Questionnaire (PASQ) scale ranging from 0 (No symptoms) to 8 (Severe, incapacitating symptoms).
Time Frame: At baseline, week 24 and week 48
Population: ITT population.
  Number of Participants Analyzed:
  Phase 1 in week 24: 3
  Phase 2 (Group A) in week 24: 13
  Phase 2 (Group B) in week 24: 69
  Phase 2 (Group C) in week 24: 25
  Phase 2 (Group A) in week 48: 13
  Phase 2 (Group B) in week 48: 68
  Phase 2 (Group C) in week 48: 26
  NA = Not Applicable
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Phase 1 Only: Lanreotide Autogel 120 mg: Only 15 subjects participated only in phase 1 and did not move on to phase 2. The other entered in phase 2 according to IGF-1 level. Subjects in phase 1 received 5 injections of Lanreotide Autogel 120 mg subcutaneously (SC) at baseline and weeks 6, 12, 18 and 24. Baseline and week 24 injections were administered in the investigational centre, whereas the patient could receive weeks 6, 12 and 18 injections at home as part of the subject's normal medical care, completing details of the injection in the diary cards provided.
Arm/Group | Phase 1 Only: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Number analyzed (Participants) | 15 | 13 | 70 | 26
Units on a scale
  Baseline - Headache | 2.73 (2.71) | 2.15 (1.72) | 1.80 (1.73) | 2.04 (2.11)
  Baseline - Excessive perspiration | 2.80 (2.93) | 1.92 (2.50) | 2.41 (2.18) | 2.08 (2.21)
  Baseline - Fatigue | 3.40 (2.85) | 4.23 (1.48) | 3.27 (2.36) | 3.31 (2.63)
  Baseline - Soft tissue swelling | 1.13 (1.77) | 2.77 (2.20) | 1.81 (2.02) | 1.42 (1.88)
  Baseline - Arthralgia | 2.73 (3.17) | 3.46 (2.30) | 3.13 (2.42) | 4.42 (2.35)
  Week 24 - Headache | 2.67 (1.53) | 1.38 (1.45) | 1.93 (1.90) | 2.04 (1.90)
  Week 24 - Excessive perspiration | 2.00 (2.00) | 2.08 (2.02) | 2.25 (2.21) | 2.64 (2.34)
  Week 24 - Fatigue | 2.33 (1.53) | 3.85 (1.86) | 3.36 (2.56) | 4.08 (2.40)
  Week 24 - Soft tissue swelling | 1.33 (1.53) | 2.46 (1.90) | 1.71 (2.17) | 1.76 (2.13)
  Week 24 - Arthralgia | 2.00 (2.65) | 3.62 (2.79) | 3.09 (2.66) | 3.68 (2.53)
  Week 48 - Headache | NA (NA) — Phase 1 was up to Week 24 only | 1.77 (1.92) | 2.32 (2.22) | 2.62 (2.08)
  Week 48 - Excessive perspiration | NA (NA) — Phase 1 was up to Week 24 only | 2.31 (2.02) | 2.50 (2.13) | 2.50 (2.40)
  Week 48 - Fatigue | NA (NA) — Phase 1 was up to Week 24 only | 3.77 (2.55) | 3.16 (2.32) | 3.92 (2.17)
  Week 48 - Soft tissue swelling | NA (NA) — Phase 1 was up to Week 24 only | 2.85 (2.08) | 2.10 (2.39) | 1.62 (2.02)
  Week 48 - Arthralgia | NA (NA) — Phase 1 was up to Week 24 only | 3.46 (2.57) | 3.60 (2.60) | 4.04 (2.24)

9. Secondary Outcome: Mean Changes From Baseline in Quality of Life Scores (AcroQoL)
Description: AcroQoL score groups 22 components: Eight physical, Seven psychological appearance and Seven psychological personal relations, adjusted to a scale of 100, where a score of 100 corresponds to the best possible QoL and 0 to the worst.
Time Frame: At weeks 24 and 48
Population: ITT population n = Number of subjects at the visit. Phase 1 only: These subjects participated only in phase 1 & did not move onto phase 2.
  Only subjects from countries having a validated translation of the AcroQoL questionnaire (The Netherlands, Denmark, Sweden, France, Greece, Poland, South Korea, Brazil, Russia, Norway and Romania) were included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase 1 Only: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks | Overall Study
Number analyzed (Participants) | 11 | 9 | 55 | 21 | 96
Units on a scale
  At week 24 (n=1, 9, 55, 21, and 86) | 21.59 (NA) — Not applicable as there is only One subject. | -2.15 (9.58) | -0.27 (11.73) | -0.84 (11.00) | -0.35 (11.43)
  At week 48 (n=0, 9, 53, 21, and 83) | NA (NA) — Phase 1 was up to Week 24 only. | 1.31 (10.67) | -1.32 (10.17) | -1.52 (10.22) | -1.08 (10.15)

10. Secondary Outcome: Mean Changes From Baseline in Quality of Life Scores (SF-36)
Description: Short Form-36 questionnaire (SF-36) score comprises eight components: Physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health on a scale of 100, where a score of 100 corresponds to the best possible QoL and 0 to the worst.
Time Frame: At weeks 24 and 48
Population: ITT population. n = Number of subjects at the visit. Phase 1 only: These 15 subjects participated only in phase 1 and did not move on to phase 2.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase 1 Only: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks | Overall Study
Number analyzed (Participants) | 15 | 13 | 70 | 26 | 124
Units on a scale
  At week 24 (n=3, 13, 70, 26, and 112) | -0.66 (39.14) | 4.91 (22.64) | 1.79 (13.54) | -2.75 (14.87) | 1.03 (15.89)
  At week 48 (n=0, 13, 68, 26, and 107) | NA (NA) — Phase 1 was up to Week 24 only. | 4.96 (20.35) | -0.61 (12.09) | -0.62 (14.76) | 0.06 (13.93)

11. Secondary Outcome: Percentage of Subjects With Normalized IGF-1 Levels (Age and Sex Adjusted), Without Any Worsening of the AcroQoL Change Score Between Inclusion and Week 48
Description: The criterion for a subject is satisfied if he had a IGF-1 level (age and sex adjusted) without any worsening of the AcroQoL change score between Inclusion and Week 48.
Time Frame: At week 48 (End of Study)
Population: MITT population. n = Number of subjects at the visit.
  Only subjects from countries having a validated translation of the AcroQoL questionnaire (The Netherlands, Denmark, Sweden, France, Greece, Poland, South Korea, Brazil, Russia, Norway and Romania) were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 85
Percentage of subjects
  Phase I / Group A (n=9) | 44.4 [12.0 to 76.9]
  Phase I / Group B (n=55) | 47.2 [33.7 to 60.6]
  Phase I / Group C (n=21) | 38.1 [17.3 to 58.9]
  Overall study (n=85) | 44.6 [33.9 to 55.3]

12. Secondary Outcome: Correlation Between the Changes From Baseline in Quality of Life (AcroQoL) With the Corresponding Changes in IGF-1 Level (Expressed as % of ULN) at Each Visit
Description: AcroQoL change from Baseline to Week 24 (48) = AcroQoL at Week 24 (48) - AcroQoL at Baseline.
  IGF-1 change from Baseline to Week 24 (48) = IGF-1 at Week 24 (48) - IGF-1 at Baseline.
  Correlation presented is a Spearman correlation (non parametric).
Time Frame: At weeks 24 and 48
Population: ITT population. n = Number of subjects at the visit.
  Only subjects from countries having a validated translation of the AcroQoL questionnaire (The Netherlands, Denmark, Sweden, France, Greece, Poland, South Korea, Brazil, Russia, Norway and Romania) were included.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Overall Study
Number analyzed (Participants) | 88
Correlation coefficient
  Week 24: Phase I / Group A (n=8) | 0.43 [-0.42 to 0.86]
  Week 24: Phase I / Group B (n=55) | -0.02 [-0.28 to 0.25]
  Week 24: Phase I / Group C (n=21) | -0.41 [-0.71 to 0.04]
  Week 24: Overall study (n=85) | -0.01 [-0.23 to 0.20]
  Week 48: Phase I / Group A (n=8) | 0.69 [-0.08 to 0.93]
  Week 48: Phase I / Group B (n=53) | -0.06 [-0.32 to 0.22]
  Week 48: Phase I / Group C (n=21) | -0.09 [-0.50 to 0.35]
  Week 48: Overall study (n=82) | -0.01 [-0.22 to 0.21]

13. Secondary Outcome: Serum Growth Hormone (GH) Levels
Time Frame: At Baseline, week 24 and week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 Only: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks | Overall Study
Number analyzed (Participants) | 15 | 13 | 70 | 26 | 124
ng/mL
  ITT - Baseline (n=15, 13, 70, 26, and 124) | 1.04 (1.02) | 0.92 (0.68) | 0.92 (1.16) | 1.08 (1.17) | 0.97 (1.09)
  ITT - Week 24 (n=3, 13, 70, 26, and 112) | 4.89 (7.42) | 0.90 (0.41) | 0.95 (0.89) | 0.67 (0.55) | 0.99 (1.42)
  ITT - Week 48 (n=0, 13, 68, 26, and 107) | NA (NA) — Phase 1 was up to week 24 | 0.69 (0.31) | 0.99 (0.99) | 0.83 (0.69) | 0.92 (0.87)
  MITT - Baseline (n=0, 13, 70, 26, and 109) | NA (NA) — Phase 1 was up to week 24 only and was not part of MITT 'NA' for Phase I only group for the MITT | 0.92 (0.68) | 0.92 (1.16) | 1.08 (1.17) | 0.96 (1.11)
  MITT - Week 24 (n=0, 13, 70, 26, and 109) | NA (NA) — Phase 1 was up to week 24 only and was not part of MITT 'NA' for Phase I only group for the MITT | 0.90 (0.41) | 0.95 (0.89) | 0.67 (0.55) | 0.88 (0.78)
  MITT - Week 48 (n=0, 13, 68, 26, and 107) | NA (NA) — Phase 1 was up to week 24 only and was not part of MITT 'NA' for Phase I only group for the MITT | 0.69 (0.31) | 0.99 (0.99) | 0.83 (0.69) | 0.92 (0.87)

14. Secondary Outcome: Percentage of Subjects With GH Level Less Than or Equal to 2.5 ng/mL
Time Frame: At weeks 24 and 48
Population: n = Number of subjects at the visit.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Overall Study: Lanreotide Autogel 120 mg injections every 6 weeks, then depending on IGF-1 results at Week 24
Arm/Group | Overall Study
Number analyzed (Participants) | 124
Percentage of subjects
  ITT: Week 24 - Phase I only (n=15) | 66.7 [13.3 to 100]
  ITT: Week 24 - Phase I / Group A (n=13) | 100.0 [100.0 to 100.0]
  ITT: Week 24 - Phase I / Group B (n=70) | 91.4 [84.9 to 98.0]
  ITT: Week 24 - Phase I / Group C (n=26) | 100.0 [100.0 to 100.0]
  ITT: Week 24 - Overall study (n=124) | 93.8 [89.3 to 98.2]
  ITT: Week 48 - Phase I / Group A (n=13) | 100.0 [100.0 to 100.0]
  ITT: Week 48 - Phase I / Group B (n=70) | 92.6 [86.4 to 98.9]
  ITT: Week 48 - Phase I / Group C (n=26) | 96.2 [88.8 to 100.0]
  ITT: Week 48 - Overall study (n=124) | 94.4 [90.0 to 98.8]
  MITT: Week 24 - Phase I / Group A (n=13) | 100.0 [100.0 to 100.0]
  MITT: Week 24 - Phase I / Group B (n=70) | 91.4 [84.9 to 98.0]
  MITT: Week 24 - Phase I / Group C (n=26) | 100.0 [100.0 to 100.0]
  MITT: Week 24 - Overall study (n=109) | 94.5 [90.2 to 98.8]
  MITT: Week 48 - Phase I / Group A (n=13) | 100.0 [100.0 to 100.0]
  MITT: Week 48 - Phase I / Group B (n=70) | 92.6 [86.4 to 98.9]
  MITT: Week 48 - Phase I / Group C (n=26) | 96.2 [88.8 to 100]
  MITT: Week 48 - Overall study (n=109) | 94.4 [90.0 to 98.8]

15. Secondary Outcome: Subject Treatment Schedule Preference
Description: At week 24, the preference assessed between Octreotide Long Acting Repeatable intramuscular injection (Oct-LAR IM) every 4 weeks and Lanreotide Autogel 120 mg subcutaneous injection (SC) every 6 weeks.
  At week 48, the preference is assessed between Oct-LAR IM every 4 weeks and Lanreotide Autogel 120 mg SC either injected every 4, 6 or 8 weeks (as injected during Phase II of the study).
Time Frame: At weeks 24 and 48
Population: ITT population. n = Number of subjects at the visit.
  Lan: Lanreotide
  W: Week
  Inj: Injection
  Wks: Weeks
  Phs: Phase
  Grp: Group
  evy: every
Measure: Number; unit: Percentage of subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 124
Percentage of subjects
  W24:Oct-LAR IM inj evy 4 wks Phs 1 only (n=15) | 20
  W24:Lan Autogel inj evy 6 wks Phs 1 only (n=15) | 80
  W24:Oct-LAR IM inj evy 4 wks Phs 1/Grp A(n=13) | 7.7
  W24:Lan Autogel inj evy 6 wks Phs 1/Grp A(n=13) | 92.3
  W24:Oct-LAR IM inj evy 4 wks Phs 1/Grp B(n=70) | 10.3
  W24:Lan Autogel inj evy 6 wks Phs 1/Grp B(n=70) | 85.3
  W24:Non precised Phs 1/Grp B (n=70) | 4.4
  W24:Oct-LAR IM inj evy 4 wks Phs 1/Grp C(n=26) | 3.8
  W24:Lan Autogel inj every 6 wks Phs 1/Grp C(n=26) | 96.2
  W 24:Oct-LAR IM inj evy 4 wks-Overall study(n=124) | 8.9
  W24:Lan Autogel inj evy 6 wks-Overall study(n=124) | 88.4
  W 24: Non precised - Overall study (n=124) | 2.7
  W48:Oct-LAR IM inj evy 4 wks Phs 1/Grp A(n=13) | 15.4
  W48:Lan Autogel inj evy 6 wks Phs 1/Grp A(n=13) | 76.9
  W48:Non precised Phs 1/Grp A (n=13) | 7.7
  W48:Oct-LAR IM inj evy 4 wks Phs 1/Grp B(n=70) | 14.7
  W48:Lan Autogel inj evy 4 wks Phs 1/Grp B(n=70) | 1.5
  W48:Lan Autogel inj evy 6 wks Phs 1/Grp B(n=70) | 77.9
  W48:Non precised Phs 1/Grp B (n=70) | 5.9
  W48:Oct-LAR IM inj evy 4 wks Phs 1/Grp C(n=26) | 7.7
  W48:Lan Autogel inj evy 8 wks Phs 1/Grp C(n=26) | 92.3
  W48:Oct-LAR IM inj evy 4 wks-Overall study(n=124) | 13.1
  W48:Lan Autogel inj evy 4 wks-Overall study(n=124) | 10.3
  W48:Lan Autogel inj evy 6 wks-Overall study(n=124) | 49.5
  W48:Lan Autogel inj evy 8 wks-Overall study(n=124) | 22.4
  W48:Non precised-Overall study (n=124) | 4.7

ADVERSE EVENTS:
Time Frame: Up to week 48
Arm/Group | Phase 1: Lanreotide Autogel 120 mg | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/13 | 4/70 | 2/26
Other Adverse Events (participants affected / at risk) | 12/15 | 10/13 | 48/70 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Lanreotide Autogel 120 mg (N=15) | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks (N=13) | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks (N=70) | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks (N=26)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Lanreotide Autogel 120 mg (N=15) | Phase 2 (Group A): Lanreotide Autogel 120 mg Every 4 Weeks (N=13) | Phase 2 (Group B): Lanreotide Autogel 120 mg Every 6 Weeks (N=70) | Phase 2 (Group C): Lanreotide Autogel 120 mg Every 8 Weeks (N=26)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (21) | 1 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (7) | 3 (3)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 6 (15) | 2 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (8) | 2 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 3 (3)
Application site pain (General disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Nodule (General disorders) | 1 (2) | 0 (0) | 1 (3) | 1 (2)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (5)
Migraine (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Podagra (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 2 (3) | 7 (7) | 4 (5)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
High density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate contr (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphangiectasia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presbyopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No